CLINICAL TRIAL: NCT00045435
Title: Nonmyeloablative Allogeneic Peripheral Blood Stem Cell Transplantation From HLA Matched Related Donors for Treatment of Older Patients With De Novo or Secondary Acute Myeloid Leukemia in First Complete Remission
Brief Title: Reduced Intensity Donor Peripheral Blood Stem Cell Transplant in Treating Patients With De Novo or Secondary Acute Myeloid Leukemia in Remission
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Brenda Sandmaier, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1654.00; NCI-2011-01307 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Results first posted 2017-03-16 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Acute Myeloid Leukemia With Multilineage Dysplasia Following Myelodysplastic Syndrome; Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Secondary Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — fludarabine phosphate; Whole-Body Irradiation; Cyclosporine; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (nonmyeloablative donor PBSC transplant) (Experimental): CONDITIONING REGIMEN: Patients receive fludarabine phosphate IV on days -4 to -2 and undergo TBI on day 0.
  TRANSPLANT: Patients undergo allogeneic PBSC transplant on day 0.
  IMMUNOSUPPRESSION: Patients receive CSP PO BID on days -3 to 56 with taper to day 77. Patients also receive MMF PO BID on days 0-27.
  Interventions: Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation; Drug: fludarabine phosphate; Radiation: total-body irradiation; Drug: cyclosporine; Drug: mycophenolate mofetil; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation — Undergo nonmyeloablative allogeneic PBSC transplant
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Radiation: total-body irradiation — Undergo TBI
  Other Names: TBI
Drug: cyclosporine — Given PO
  Other Names: ciclosporin; cyclosporin; cyclosporin A; CYSP; Sandimmune
Drug: mycophenolate mofetil — Given PO
  Other Names: Cellcept; MMF
Procedure: peripheral blood stem cell transplantation — Undergo nonmyeloablative allogeneic PBSC transplant
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell

SUMMARY:
This phase II trial studies how well reduced intensity donor peripheral blood stem cell (PBSC) transplant works in treating patients with de novo or secondary acute myeloid leukemia (AML) in remission. Giving low doses of chemotherapy, such as fludarabine phosphate, and total-body irradiation (TBI) before a donor PBSC transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving cyclosporine and mycophenolate mofetil after the transplant may stop this from happening

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if a one-year disease free survival of >= 35% can be achieved among patients >= 55 years old with de novo and secondary AML in first complete remission (CR1) who undergo nonmyeloablative hematopoietic stem cell transplant (HSCT) from human leukocyte antigen (HLA) identical related donors.

II. To determine if a day +200 nonrelapse related mortality of < 15% can be achieved among patients >= 55 years old with de novo and secondary AML in CR1 who undergo nonmyeloablative HSCT from HLA identical related donors.

OUTLINE:

CONDITIONING REGIMEN: Patients receive fludarabine phosphate intravenously (IV) on days -4 to -2 and undergo TBI on day 0.

TRANSPLANT: Patients undergo allogeneic PBSC transplant on day 0.

IMMUNOSUPPRESSION: Patients receive cyclosporine (CSP) orally (PO) twice daily (BID) on days -3 to 56 with taper to day 77. Patients also receive mycophenolate mofetil (MMF) PO BID on days 0-27.

After completion of study treatment, patients are followed up on days 28, 56, and 84; months 6, 12, 18, and 24; and then yearly for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with de novo AML (French-American-British [FAB] MO-M2, M4-M7) or secondary AML who achieve CR1 after induction chemotherapy and one or two cycles of consolidation chemotherapy
* Transplant conditioning must occur within 6 months of diagnosis
* Patient enrollment must be approved by the Fred Hutchinson Cancer Research Center (FHCRC) principal investigator (PI) or the PI's designee
* DONOR: Related donor who is genotypically or phenotypically identical
* DONOR: Age >= 12 years
* DONOR: Donor must consent to filgrastim (G-CSF) administration and leukapheresis
* DONOR: Donor must have adequate veins for leukapheresis or agree to placement of central venous catheter (femoral, subclavian)

Exclusion Criteria:

* AML FAB M3
* AML involvement of the central nervous system (CNS) as defined by a positive cytospin of cerebral spinal fluid at the time of enrollment
* Presence of circulating leukemic blasts (in the peripheral blood) detected by standard pathology
* Human immunodeficiency virus (HIV) seropositivity
* Fungal infections with radiographic progression after receipt of amphotericin B or active triazole for greater than one month
* Diffusion capacity of carbon monoxide (DLCO) corrected < 40%
* Total lung capacity (TLC) < 40%
* Forced expiratory volume in one second (FEV1) < 40% or requiring supplementary oxygen
* The FHCRC principal investigator of the study must approve enrollment of all patients with pulmonary nodules
* Cardiac ejection fraction < 40%
* Patients with clinical or laboratory evidence of liver disease would be evaluated for the cause of liver disease, its clinical severity in terms of liver function, bridging fibrosis, and the degree of portal hypertension; patients will be excluded if they are found to have fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction evinced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3mg/dL, or symptomatic biliary disease
* Karnofsky Performance Score < 70
* Fertile men or women unwilling to use contraceptive techniques during and for 12 months following treatment
* Females who are pregnant or breastfeeding
* No intensive chemotherapy can be given within three weeks (or the interval in which a cycle of standard chemotherapy would be administered in a non-transplant setting) prior to initiating the nonmyeloablative transplant conditioning
* Patients with active non-hematologic malignancies (except non-melanoma skin cancers)
* Patients with a history of non-hematologic malignancies (except non-melanoma skin cancers) currently in a complete remission, who are less than 5 years from the time of complete remission, and have a > 20% risk of disease recurrence
* Patients with active bacterial or fungal infections unresponsive to medical therapy
* DONOR: Identical twin
* DONOR: Pregnancy
* DONOR: HIV seropositivity
* DONOR: Inability to achieve adequate venous access
* DONOR: Known allergy to G-CSF
* DONOR: Current serious systemic illness

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2002-04 (Actual); Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Sandmaier, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - OHSU Cancer Institute, Portland, Oregon
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington

REFERENCES:
- [Derived] Cooper JP, Storer BE, Granot N, Gyurkocza B, Sorror ML, Chauncey TR, Shizuru J, Franke GN, Maris MB, Boyer M, Bruno B, Sahebi F, Langston AA, Hari P, Agura ED, Lykke Petersen S, Maziarz RT, Bethge W, Asch J, Gutman JA, Olesen G, Yeager AM, Hubel K, Hogan WJ, Maloney DG, Mielcarek M, Martin PJ, Flowers MED, Georges GE, Woolfrey AE, Deeg JH, Scott BL, McDonald GB, Storb R, Sandmaier BM. Allogeneic hematopoietic cell transplantation with non-myeloablative conditioning for patients with hematologic malignancies: Improved outcomes over two decades. Haematologica. 2021 Jun 1;106(6):1599-1607. doi: 10.3324/haematol.2020.248187. PMID 32499241

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Nonmyeloablative Donor PBSC Transplant): Patients receive fludarabine phosphate IV on days -4 to -2 and undergo TBI & allogeneic PBSC transplant on day 0. Patients also receive CSP PO BID on days -3 to 56 with taper to day 77, and MMF PO BID on days 0-27.
  Nonmyeloablative allogeneic hematopoietic stem cell transplantation: Undergo nonmyeloablative allogeneic peripheral blood stem cell transplant
  Fludarabine phosphate: Given IV
  Total-body irradiation: Undergo total-body irradiation
  Cyclosporine: Given PO
  Mycophenolate mofetil: Given PO
  Peripheral blood stem cell transplantation: Undergo nonmyeloablative allogeneic peripheral blood stem cell transplant
Period: Overall Study
Arm/Group | Treatment (Nonmyeloablative Donor PBSC Transplant)
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Nonmyeloablative Donor PBSC Transplant)
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 7
Age, Continuous [Median (Full Range); unit: years] | 64.8 [56 to 72.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival-incidence of Survival Without Relapse
Description: Sufficient evidence will be taken to be an observed rate of DFS at one year after transplant that corresponds to a one-sided 95% confidence interval with an upper limit lower than 35%.
Time Frame: By 1 year after transplant
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Nonmyeloablative Donor PBSC Transplant)
Number analyzed (Participants) | 17
percentage of participants | 47
Statistical Analysis 1: Comparison: Treatment (Nonmyeloablative Donor PBSC Transplant); The study was to be stopped after 20 patients if the upper bound of a 1-sided 95% confidence interval for relapse-free survival was <35%; Test type: Other; Percent = 47, 95% CI 1-sided [upper limit 69] — The criterion for stopping was not met

2. Primary Outcome: Nonrelapse Mortality (NRM)-Incidence of Nonrelapse Death
Description: Defined as death without morphologic evidence of disease. Sufficient evidence will be taken to be an observed rate of NRM within 200 days of transplant that corresponds to a one-sided 80% confidence interval with a lower limit greater than 15%.
Time Frame: 200 days after transplant
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Nonmyeloablative Donor PBSC Transplant)
Number analyzed (Participants) | 17
percentage of participants | 6
Statistical Analysis 1: Comparison: Treatment (Nonmyeloablative Donor PBSC Transplant); The study was to be stopped if the lower bound of a 1-sided 80% confidence interval for NRM was greater than 15%; Test type: Other; percent = 6, 80% CI 1-sided [lower limit 1] — The stopping criterion was not met

3. Secondary Outcome: Overall Survival
Description: Percent patients surviving.
Time Frame: By 1 year after transplant
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Nonmyeloablative Donor PBSC Transplant)
Number analyzed (Participants) | 17
percentage of participants | 70.6

4. Secondary Outcome: Incidence of Relapse
Description: Percent patients with relapsed disease post-transplant.
Time Frame: By 1 year after transplant
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Nonmyeloablative Donor PBSC Transplant)
Number analyzed (Participants) | 17
percentage of participants | 41.2

5. Secondary Outcome: Incidence of Rejection
Description: Percent patients who developed infections post-transplant.
Time Frame: By 1 year after transplant
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Nonmyeloablative Donor PBSC Transplant)
Number analyzed (Participants) | 17
percentage of participants | 0

6. Secondary Outcome: Incidence of Acute and Chronic GVHD
Description: Percent patients with acute/chronic GVHD
Time Frame: aGVHD: 100 days after transplant; cGVHD: 1 Year after transplant.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Nonmyeloablative Donor PBSC Transplant)
Number analyzed (Participants) | 17
percentage of participants
  Grade II-IV aGVHD | 35.3
  cGVHD | 35.3

ADVERSE EVENTS:
Time Frame: AEs: Conditioning through Day 100; SAEs: Conditioning through Day 200
Arm/Group | Treatment (Nonmyeloablative Donor PBSC Transplant)
Serious Adverse Events (participants affected / at risk) | 5/17
Other Adverse Events (participants affected / at risk) | 4/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nonmyeloablative Donor PBSC Transplant) (N=17)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
GVHD (Immune system disorders) | 1 (1)
Secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nonmyeloablative Donor PBSC Transplant) (N=17)
Heart failure (Cardiac disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Neutrophil count decreased (Investigations) | 2 (2)
Thromboembolic event (Vascular disorders) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes